CLINICAL TRIAL: NCT03083210
Title: PILOT STUDY OF LANREOTIDE IN METASTATIC OR RECURRENT GRADE I-II HINDGUT NET
Brief Title: Study of Lanreotide in Metastatic or Recurrent Grade I-II Hindgut NET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-11-017
Record Dates: First submitted 2017-02-15; First posted 2017-03-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide

STUDY DESIGN:
Intervention Model Description: Lanreotide, at a dose of 120mg subcutaneous injection every 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lanreotide (Experimental): Lanreotide, at a dose of 120mg will be administered without dose adjustment, by means of deep subcutaneous injection every 28 days.
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide — Lanreotide, at a dose of 120mg subcutaneous injection every 28 days.

SUMMARY:
Clinical data from uncontrolled retrospective or prospective studies have initially demonstrated antiproliferative effects of lanreotide in limited number of patients lanreotide Autogel® has recently been approved in more than 40 countries for the treatment of GEP-NET patients, this is based on the results of CLARINET study, the largest prospective trial to evaluate the antiproliferative effects of lanreotide Autogel® in subjects with nonfunctional GEP-NETs. The study enrolled 204 subjects (101 subjects were randomized to lanreotide Autogel® group and 103 subjects were randomized to placebo group, came from 14 countries) with well or moderately differentiated non-functioning GEP-NETs, including pancreatic and gastrointestinal tumors, and defined as having less than 10% of proliferation marker Ki67. The study had shown that treatment with lanreotide Autogel® significantly prolonged progression-free survival in subjects with GEP-NETs compared to treatment with placebo in the primary analysis (median progression-free survival, not reached vs. 18.0 months, P< 0.001 by the stratified log-rank test; hazard ratio for progression or death with lanreotide vs. placebo, 0.47; 95% confidence interval (CI), 0.30 to 0.73) [5].

The indication of GEP-NETs granted for lanreotide Autogel® in the USA is for the treatment of patients with unresectable, well or moderately differentiated, locally advanced or metastatic gastroenteropancreatic neuroendocrine tumors (GEP-NETs) to improve progression-free survival; and in the European Union (EU) is for treatment of grade 1 and a subset of grade 2 (Ki67 index up to 10%) gastroenteropancreatic neuroendocrine tumors of midgut, pancreatic or unknown origin where hindgut sites of origin have been excluded, in adult patients with unresectable locally advanced or metastatic disease. The addition of an indication for the treatment of patients with GEP-NETs has been approved by more than 15 other authorities including in Canada, Australia and some Asian countries, etc.

DETAILED DESCRIPTION:
Patients with advanced hindgut NET who don't receive prior systemic therapies will receive laneotide. Study-arm is composed of 28 patients. Laneotide 120mg s.c. once every a 28 day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed well differentiated or moderate differentiated neuroendocrine tumor. WHO 2010 Grade 1 or 2
* Age >20
* Measurable disease by RECIST v 1.0
* Primary tumor were located in hindgut, colorectal areas.
* Non functioning or functioning NETs
* Unresectable locally advanced or metastatic disease

Exclusion Criteria:

* Prior receiving systemic therapies including interferon, chemotherapy, PRRT, chemoembolization or a somatostatin analogue at any time (unless they had received it >6 months previously and for <15 days).
* Multiple endocrine neoplasia
* Previous cancer except in the case of patients with treated or untreated in situ cervical or uterine carcinoma or basal cell skin cancer or patients with other cancers who had been treated with curative intent and had been disease free for > 5 years
* Foregut, midgut, and pancreatic NETs and NETs of unknown primary origin Cross reference: Hindgut: Distal 1/3rd transverse colon, descending colon, sigmoid colon, rectum, upper anal canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Youngsuk Park, Seoul, South Korea